CLINICAL TRIAL: NCT03143153
Title: A Randomized Phase 3 Study of Nivolumab Plus Ipilimumab or Nivolumab Combined With Fluorouracil Plus Cisplatin Versus Fluorouracil Plus Cisplatin in Subjects With Unresectable Advanced, Recurrent or Metastatic Previously Untreated Esophageal Squamous Cell Carcinoma
Brief Title: A Study to Evaluate Efficacy in Subjects With Esophageal Cancer Treated With Nivolumab and Ipilimumab or Nivolumab Combined With Fluorouracil Plus Cisplatin Versus Fluorouracil Plus Cisplatin
Acronym: CheckMate 648
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-648; 2016-001514-20 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab + Ipilimumab (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab + Cisplatin + Fluorouacil (Experimental)
  Interventions: Biological: Nivolumab; Drug: Cisplatin; Drug: Fluorouracil
- Cisplatin + Fluorouracil (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Fluorouracil

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558 (Nivolumab); Opdivo (Nivolumab)
  Arms: Nivolumab + Cisplatin + Fluorouacil; Nivolumab + Ipilimumab
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016 (Ipilimumab); Yervoy (Ipilimumab)
  Arms: Nivolumab + Ipilimumab
Drug: Cisplatin — Specified dose on specified days
  Arms: Cisplatin + Fluorouracil; Nivolumab + Cisplatin + Fluorouacil
Drug: Fluorouracil — Specified dose on specified days
  Arms: Cisplatin + Fluorouracil; Nivolumab + Cisplatin + Fluorouacil

SUMMARY:
The main purpose of this study is to compare how long subjects with esophageal cancer live overall or live without disease progression after receiving nivolumab and ipilimumab or nivolumab combined with fluorouracil plus cisplatin versus fluorouracil plus cisplatin

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed squamous cell carcinoma or adenosquamous cell carcinoma of esophagus
* Male or Female at least 18 years of age
* Must have esophageal cancer that cannot be operated on, or treated with definitive chemoradiation with curative intent, that is advanced, reoccurring or has spread out
* Must have full activity or, if limited, must be able to walk and carry out light activities such as light house work or office work
* Must agree to provide tumor tissue sample, either from a previous surgery or biopsy within 6 months or fresh, prior to the start of treatment in this study

Exclusion Criteria

* Presence of tumor cells in the brain or spinal cord which are symptomatic or require treatment
* Active known or suspected autoimmune disease
* Any serious or uncontrolled medical disorder or active infection
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any positive test result for hepatitis B or C indicating acute or chronic infection and/or detectable virus

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (190):
- United States (16):
  - Local Institution - 0191, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Local Institution - 0188, Denver, Colorado
  - University Of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Local Institution - 0186, Miami, Florida
  - Local Institution - 0225, Tampa, Florida
  - Local Institution - 0074, Atlanta, Georgia
  - Local Institution - 0032, Marietta, Georgia
  - Hackensack Meridian Jersey Shore University Medical Center, Neptune City, New Jersey
  - Oncology Associates Of Oregon, Pc, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Local Institution - 0210, Dallas, Texas
  - Local Institution - 0028, Houston, Texas
  - Local Institution - 0190, Roanoke, Virginia
  - Local Institution - 0203, Morgantown, West Virginia
- Argentina (4):
  - Local Institution - 0050, Capital Federal, Buenos Aires
  - Local Institution - 0086, Rosario, Santa Fe Province
  - Local Institution - 0048, Buenos Aires
  - Local Institution - 0087, La Rioja
- Australia (3):
  - Local Institution - 0232, Tamworth, New South Wales
  - Local Institution - 0011, Douglas, Queensland
  - Local Institution - 0010, Murdoch, Western Australia
- Local Institution - 0241, Salzburg, Austria
- Brazil (9):
  - Local Institution - 0017, Salvador, Estado de Bahia
  - Local Institution - 0227, Ipatinga, Minas Gerais
  - Local Institution - 0021, Ijuí, Rio Grande do Sul
  - Local Institution - 0016, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0019, Barretos, São Paulo
  - Local Institution - 0226, Jaú, São Paulo
  - Local Institution - 0018, São José do Rio Preto, São Paulo
  - Local Institution - 0228, Rio de Janeiro
  - Local Institution - 0020, São Paulo
- Canada (4):
  - Local Institution - 0095, Moncton, New Brunswick
  - Local Institution - 0082, Montreal, Quebec
  - Local Institution - 0222, Montreal, Quebec
  - Local Institution - 0037, Trois-Rivières, Quebec
- Chile (2):
  - Local Institution - 0053, Santiago, Santiago Metropolitan
  - Local Institution - 0214, Santiago, Santiago Metropolitan
- China (23):
  - Local Institution - 0207, Hefei, Anhui
  - Local Institution - 0197, Hefei, Anhui
  - Local Institution - 0182, Beijing, Beijing Municipality
  - Local Institution - 0179, Beijing, Beijing Municipality
  - Local Institution - 0216, Beijing, Beijing Municipality
  - Local Institution - 0217, Fuzhou, Fujian
  - Local Institution - 0219, Fuzhou, Fujian
  - Local Institution - 0199, Shantou, Guangdong
  - Local Institution - 0185, Harbin, Heilongjiang
  - Local Institution - 0193, Zhengzhou, Henan
  - Local Institution - 0195, Zhengzhou, Henan
  - Local Institution - 0194, Zhengzhou, Henan
  - Local Institution - 0249, Changsha, Hunan
  - Local Institution - 0212, Changsha, Hunan
  - Local Institution - 0201, Nanjing, Jiangsu
  - Local Institution - 0180, Changchun, Jilin
  - Local Institution - 0183, Xi'an, Shan3xi
  - Local Institution - 0215, Shanghai, Shanghai Municipality
  - Local Institution - 0200, Shanghai, Shanghai Municipality
  - Local Institution - 0184, Hangzhou, Zhejiang
  - Local Institution - 0247, Linhai, Zhejiang
  - Local Institution - 0220, Shenyang
  - Local Institution - 0248, Xi'an
- Colombia (4):
  - Local Institution - 0059, Bogotá
  - Local Institution - 0058, Medellín
  - Local Institution - 0224, Montería
  - Local Institution - 0094, Pereira
- Czechia (3):
  - Local Institution - 0083, Brno
  - Local Institution - 0008, Brno
  - Local Institution - 0006, Nový Jičín
- Local Institution - 0099, Odense, Denmark
- France (6):
  - Local Institution - 0116, Lille, Nord
  - Local Institution - 0114, Caen
  - Local Institution - 0112, Montpellier
  - Local Institution - 0113, Rennes
  - Local Institution - 0242, Toulouse
  - Local Institution - 0115, Villejuif
- Hong Kong (2):
  - Local Institution - 0035, Hong Kong
  - Local Institution - 0070, Kowloon
- Italy (4):
  - Local Institution - 0085, Bergamo
  - Local Institution - 0039, Milan
  - Local Institution - 0084, Padua
  - Local Institution - 0240, Pisa
- Japan (54):
  - Local Institution - 0152, Akita, Akita
  - Local Institution - 0104, Hirosaki-shi, Aomori
  - Local Institution - 0173, Kashiwa-shi, Chiba
  - Local Institution - 0169, Matsuyama, Ehime
  - Local Institution - 0119, Matsuyama, Ehime
  - Local Institution - 0174, Fukuoka, Fukuoka
  - Local Institution - 0142, Fukuoka, Fukuoka
  - Local Institution - 0103, Fukushima, Fukushima
  - Local Institution - 0154, Gifu, Gifu
  - Local Institution - 0176, Ōta, Gunma
  - Local Institution - 0100, Hiroshima, Hiroshima
  - Local Institution - 0111, Sapporo, Hokkaido
  - Local Institution - 0170, Akashi-shi, Hyōgo
  - Local Institution - 0172, Kobe, Hyōgo
  - Local Institution - 0118, Kobe, Hyōgo
  - Local Institution - 0171, Kanazawa, Ishikawa-ken
  - Local Institution - 0229, Kagoshima, Kagoshima-ken
  - Local Institution - 0127, Isehara, Kanagawa
  - Local Institution - 0109, Kawasaki-shi, Kanagawa
  - Local Institution - 0105, Sagamihara-shi, Kanagawa
  - Local Institution - 0147, Yokohama, Kanagawa
  - Local Institution - 0117, Yokohama, Kanagawa
  - Local Institution - 0141, Kumamoto, Kumamoto
  - Local Institution - 0120, Kamigyō-ku, Kyoto
  - Local Institution - 0144, Sendai, Miyagi
  - Local Institution - 0146, Niigata, Niigata
  - Local Institution - 0135, Kurashiki-shi, Okayama-ken
  - Local Institution - 0137, Okayama, Okayama-ken
  - Local Institution - 0221, Hirakata, Osaka
  - Local Institution - 0138, Osaka, Osaka
  - Local Institution - 0098, Sayama, Osaka
  - Local Institution - 0107, Suita, Osaka
  - Local Institution - 0139, Takatsuki, Osaka
  - Local Institution - 0230, Hidaka-shi, Saitama
  - Local Institution - 0175, Kitaadachi-gun, Saitama
  - Local Institution - 0143, Sunto-gun, Shizuoka
  - Local Institution - 0148, Shimotsuga-gun, Tochigi
  - Local Institution - 0106, Bunkyo-ku, Tokyo
  - Local Institution - 0110, Bunkyo-ku, Tokyo
  - Local Institution - 0136, Chuo-ku, Tokyo
  - Local Institution - 0128, Chuo-ku, Tokyo
  - Local Institution - 0126, Koto-ku, Tokyo
  - Local Institution - 0156, Minato-ku, Tokyo
  - Local Institution - 0245, Ōta-ku, Tokyo
  - Local Institution - 0140, Shinagawa-ku, Tokyo
  - Local Institution - 0196, Shinjuku-Ku, Tokyo
  - Local Institution - 0155, Shinjuku-ku, Tokyo
  - Local Institution - 0231, Toyama, Toyama
  - Local Institution - 0178, Wakayama, Wakayama
  - Local Institution - 0238, Ube-shi, Yamaguchi
  - Local Institution - 0101, Chiba
  - Local Institution - 0153, Chiba
  - Local Institution - 0145, Kyoto
  - Local Institution - 0108, Shizuoka
- Mexico (4):
  - Local Institution - 0090, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 0102, Mexico City, Mexico City
  - Local Institution - 0071, Mérida, Yucatán
  - Local Institution - 0234, San Luis Potosí City
- Peru (3):
  - Local Institution - 0092, Callao
  - Local Institution - 0060, Lima
  - Local Institution - 0093, Lima
- Poland (2):
  - Local Institution - 0024, Lublin
  - Local Institution - 0022, Warsaw
- Local Institution - 0243, Porto, Portugal
- Romania (4):
  - Local Institution - 0081, Bucharest
  - Local Institution - 0079, Cluj-Napoca
  - Local Institution - 0076, Craiova
  - Local Institution - 0080, Suceava
- Russia (2):
  - Local Institution - 0089, Moscow
  - Local Institution - 0088, Saint Petersburg
- Singapore (2):
  - Local Institution - 0033, Singapore, Central Singapore
  - Local Institution - 0034, Singapore
- South Korea (14):
  - Local Institution - 0129, Seongnam-si, Kyǒnggi-do
  - Local Institution - 0165, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0166, Busan
  - Local Institution - 0150, Daegu
  - Local Institution - 0149, Daejeon
  - Local Institution - 0236, Jeonju
  - Local Institution - 0235, Seoul
  - Local Institution - 0130, Seoul
  - Local Institution - 0177, Seoul
  - Local Institution - 0168, Seoul
  - Local Institution - 0151, Seoul
  - Local Institution - 0131, Seoul
  - Local Institution - 0123, Seoul
  - Local Institution - 0157, Ulsan
- Spain (2):
  - Local Institution - 0063, Barcelona
  - Local Institution - 0062, Madrid
- Taiwan (12):
  - Local Institution - 0158, Changhua County, Changhua
  - Local Institution - 0161, Tainan, TNN
  - Local Institution - 0167, Kaohsiung City
  - Local Institution - 0133, Kaohsiung City
  - Local Institution - 0163, Kaohsiung County
  - Local Institution - 0164, Keelung
  - Local Institution - 0132, Taichung
  - Local Institution - 0160, Tainan
  - Local Institution - 0124, Taipei
  - Local Institution - 0162, Taipei
  - Local Institution - 0134, Taipei
  - Local Institution - 0159, Taoyuan District
- Turkey (Türkiye) (3):
  - Local Institution - 0096, Ankara
  - Local Institution - 0125, Diyarbakır
  - Local Institution - 0122, Edrine
- United Kingdom (5):
  - Local Institution - 0069, London, Greater London
  - Local Institution - 0066, London, Greater London
  - Local Institution - 0031, Manchester, Greater Manchester
  - Local Institution - 0237, London
  - Local Institution - 0029, Surrey

REFERENCES:
- [Derived] Zhang Y, Li C, Du K, Pengkhun N, Huang Z, Gong M, Li Y, Liu X, Li L, Wang D, Wang C, Chen F, Li J. Comparative analysis of immune checkpoint inhibitors in first-line treatment of esophageal squamous cell carcinoma: a network meta-analysis. Immunotherapy. 2023 Jul;15(10):737-750. doi: 10.2217/imt-2022-0236. Epub 2023 May 4. PMID 37139963
- [Derived] Kato K, Doki Y, Ogata T, Motoyama S, Kawakami H, Ueno M, Kojima T, Shirakawa Y, Okada M, Ishihara R, Kubota Y, Amaya-Chanaga C, Chen T, Matsumura Y, Kitagawa Y. First-line nivolumab plus ipilimumab or chemotherapy versus chemotherapy alone in advanced esophageal squamous cell carcinoma: a Japanese subgroup analysis of open-label, phase 3 trial (CheckMate 648/ONO-4538-50). Esophagus. 2023 Apr;20(2):291-301. doi: 10.1007/s10388-022-00970-1. Epub 2022 Nov 19. PMID 36401133
- [Derived] Doki Y, Ajani JA, Kato K, Xu J, Wyrwicz L, Motoyama S, Ogata T, Kawakami H, Hsu CH, Adenis A, El Hajbi F, Di Bartolomeo M, Braghiroli MI, Holtved E, Ostoich SA, Kim HR, Ueno M, Mansoor W, Yang WC, Liu T, Bridgewater J, Makino T, Xynos I, Liu X, Lei M, Kondo K, Patel A, Gricar J, Chau I, Kitagawa Y; CheckMate 648 Trial Investigators. Nivolumab Combination Therapy in Advanced Esophageal Squamous-Cell Carcinoma. N Engl J Med. 2022 Feb 3;386(5):449-462. doi: 10.1056/NEJMoa2111380. PMID 35108470
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 970 participants randomized, 936 treated.
Groups:
- Arm A: Nivolumab + Ipilimumab: Participants will receive treatment with nivolumab 3 mg/kg as a 30-minute infusion every 2 weeks and ipilimumab as a 30-minute infusion 1 mg/kg every 6 weeks.
- Arm B: Nivolumab + Chemotherapy: Participants will receive treatment with nivolumab 240 mg as a 30-minute infusion on Day 1 and Day 15, fluorouracil 800 mg/m²/day as an IV continuous infusion on Day 1 through Day 5 (for 5 days), and cisplatin 80 mg/m² as a 30- to 120-minute infusion on Day 1 of 4-week cycle.
- Arm C: Chemotherapy: Participants will receive treatment with fluorouracil 800 mg/m²/day as an IV continuous infusion from Day 1 through Day 5 (for 5 days), and cisplatin 80 mg/m² as a 30- to 120-minute infusion on Day 1 of 4-week cycle.
Period: Pre-Treatment
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Started (Started=Randomized) | 325 | 321 | 324
Completed (Completed=Treated) | 322 | 310 | 304
Not Completed | 3 | 11 | 20
Not completed — Participant request to discontinue study treatment | 0 | 0 | 2
Not completed — Participant withdrew consent | 0 | 1 | 12
Not completed — Participant no longer meets study criteria | 0 | 4 | 2
Not completed — Other Reasons | 1 | 2 | 1
Not completed — Disease Progression | 1 | 1 | 2
Not completed — Adverse event unrelated to study drug | 1 | 3 | 1
Period: Treatment
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Started | 322 | 310 | 304
Completed (Completed=continuing treatment) | 21 | 25 | 4
Not Completed | 301 | 285 | 300
Not completed — Disease progression | 174 | 184 | 193
Not completed — Study drug toxicity | 59 | 33 | 40
Not completed — Death | 5 | 3 | 4
Not completed — Adverse event unrelated to study drug | 19 | 28 | 12
Not completed — Participant request to discontinue study treatment | 13 | 15 | 20
Not completed — Participant withdrew consent | 3 | 4 | 12
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Maximum clinical benefit | 1 | 3 | 4
Not completed — Completed treatment as per Protocol | 13 | 8 | 0
Not completed — Other reasons | 12 | 7 | 15
Not completed — Not reported | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy | Total
Number analyzed (Participants) | 325 | 321 | 324 | 970
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.1) | 63.1 (9.2) | 63.3 (8.7) | 62.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 68 | 49 | 173
  Male | 269 | 253 | 275 | 797
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 79 | 85 | 84 | 248
  Black or African American | 4 | 1 | 6 | 11
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian Indian | 1 | 4 | 3 | 8
  Chinese | 71 | 74 | 70 | 215
  Japanese | 131 | 126 | 137 | 394
  Asian Other | 28 | 23 | 17 | 68
  Other | 10 | 6 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Tumor Cell PD-L1
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS will be censored on the last date the subject was known to be alive.
Time Frame: From the date of randomization to up to the date of death (up to approximately 20 months)
Population: All randomized PD-L1 expressing participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Number analyzed (Participants) | 158 | 158 | 157
Months | 13.70 [11.24 to 17.02] | 15.44 [11.93 to 19.52] | 9.07 [7.69 to 9.95]
Statistical Analysis 1: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.0010, Log Rank — Log-rank test stratified by ECOG Performance Status (0 vs 1), number of organs with metastases (<= 1 vs. >= 2) as recorded in IRT; Hazard Ratio (HR) = 0.64, 98.6% CI 2-sided [0.46 to 0.90] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.0010, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.49 to 0.84] — Stratified Cox proportional hazard model
Statistical Analysis 3: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.54, 99.5% CI 2-sided [0.37 to 0.80] — Stratified Cox proportional hazard model
Statistical Analysis 4: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.41 to 0.71] — Stratified Cox proportional hazard model

2. Primary Outcome: Progression-free Survival (PFS) as Assessed by BICR in Participants With Tumor Cell PD-L1
Description: Progression-free survival (PFS) is defined as the time from randomization to the date of the first documented progressive disease (PD) per Blinded Independent Central Review (BICR) or death due to any cause. Participants who die without a reported prior PD per BICR (and die without start of subsequent therapy) will be considered to have progressed on the date of death. Participants who did not have documented PD per BICR per RECIST1.1 criteria and who did not die, will be censored at the date of the last evaluable tumor assessment on or prior to initiation of the subsequent anti-cancer therapy. Participants who did not have any on-study tumor assessments and did not die (or died after initiation of the subsequent anti-cancer therapy) will be censored at the randomization date. Participants who started any subsequent anti-cancer therapy without a prior reported PD per BICR will be censored at the last tumor assessment on or prior to initiation of the subsequent anti-cancer therapy.
Time Frame: From the date of randomization to up to the date of the first documented disease progression or death (up to approximately 9 months)
Population: All randomized PD-L1 expressing participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Number analyzed (Participants) | 158 | 158 | 157
Months | 4.04 [2.40 to 4.93] | 6.93 [5.68 to 8.34] | 4.44 [2.89 to 5.82]
Statistical Analysis 1: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.8958, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 98.5% CI 2-sided [0.73 to 1.43] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.8958, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.78 to 1.34] — Stratified Cox proportional hazard model
Statistical Analysis 3: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0023, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 98.5% CI 2-sided [0.46 to 0.92] — Stratified Cox proportional hazard model
Statistical Analysis 4: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0023, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.86] — Stratified Cox proportional hazard model

3. Secondary Outcome: Overall Survival (OS) in All Randomized Participants
Description: as for outcome 1
Time Frame: From the date of randomization to up to the date of death (up to approximately 16 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Number analyzed (Participants) | 325 | 321 | 324
Months | 12.75 [11.27 to 15.47] | 13.21 [11.14 to 15.70] | 10.71 [9.40 to 11.93]
Statistical Analysis 1: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.0110, Log Rank — Log-rank test stratified by ECOG Performance Status (0 vs 1), number of organs with metastases (<= 1 vs. >= 2), PD-L1 status (>= 1% vs. < 1% or indeterminate) as recorded in IRT; Hazard Ratio (HR) = 0.78, 95% CI [0.65 to 0.95] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; p = 0.0110, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.78, 98.2% CI [0.62 to 0.98] — Stratified Cox proportional hazard model
Statistical Analysis 3: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0021, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.74, 99.1% CI [0.58 to 0.96] — Stratified Cox proportional hazard model
Statistical Analysis 4: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0021, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.61 to 0.90] — Stratified Cox proportional hazard model

4. Secondary Outcome: Progression-free Survival (PFS) in All Randomized Participants as Assessed by BICR
Description: as for outcome 2
Time Frame: From the date of randomization to up to the date of the first documented disease progression or death (up to approximately 7 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Number analyzed (Participants) | 325 | 321 | 324
Months | 2.92 [2.66 to 4.17] | 5.82 [5.55 to 7.00] | 5.59 [4.27 to 5.88]
Statistical Analysis 1: Comparison: Arm A: Nivolumab + Ipilimumab vs Arm C: Chemotherapy; Hazard Ratio is Arm A: Nivolumab + Ipilimumab over Arm C: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [1.04 to 1.52] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0355, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 0.99] — Stratified Cox proportional hazard model
Statistical Analysis 3: Comparison: Arm B: Nivolumab + Chemotherapy vs Arm C: Chemotherapy; Hazard Ratio is Arm B: Nivolumab + Chemotherapy over Arm C: Chemotherapy; Test type: Superiority; p = 0.0355, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.81, 98.5% CI 2-sided [0.64 to 1.04] — Stratified Cox proportional hazard model

5. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BICR
Description: Objective response rate (ORR) is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). Best overall response (BOR) is defined as the best response designation as determined by BICR, recorded between the date of randomization and the date of objectively documented progression (per RECIST 1.1) or the date of subsequent anti-cancer therapy (including tumor-directed radiotherapy and tumor-directed surgery), whichever occurs first. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions. Complete response is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Time Frame: From the date of randomization to up to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (up to 40 months)
Population: All randomized PD-L1 expressing participants and all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Chemotherapy | Arm C: Chemotherapy
Number analyzed (Participants) | 325 | 321 | 324
Percentage of participants
  Participants with baseline PD-L1 status < 1%: number analyzed (Participants) | 164 | 163 | 166
  Participants with baseline PD-L1 status < 1% | 20.1 [14.3 to 27.1] | 41.7 [34.1 to 49.7] | 33.7 [26.6 to 41.5]
  Participants with baseline PD-L1 status >= 1%: number analyzed (Participants) | 158 | 158 | 156
  Participants with baseline PD-L1 status >= 1% | 35.4 [28.0 to 43.4] | 53.2 [45.1 to 61.1] | 19.9 [13.9 to 27.0]
  Participants with baseline PD-L1 status < 5%: number analyzed (Participants) | 202 | 201 | 207
  Participants with baseline PD-L1 status < 5% | 22.3 [16.7 to 28.6] | 44.8 [37.8 to 51.9] | 30.9 [24.7 to 37.7]
  Participants with baseline PD-L1 status >= 5%: number analyzed (Participants) | 120 | 120 | 115
  Participants with baseline PD-L1 status >= 5% | 36.7 [28.1 to 45.9] | 51.7 [42.4 to 60.9] | 20.0 [13.1 to 28.5]
  Participants with baseline PD-L1 status < 10%: number analyzed (Participants) | 219 | 219 | 225
  Participants with baseline PD-L1 status < 10% | 23.3 [17.9 to 29.5] | 46.1 [39.4 to 53.0] | 29.3 [23.5 to 35.8]
  Participants with baseline PD-L1 status >= 10%: number analyzed (Participants) | 103 | 102 | 97
  Participants with baseline PD-L1 status >= 10% | 36.9 [27.6 to 47.0] | 50.0 [39.9 to 60.1] | 21.6 [13.9 to 31.2]
  Participants with baseline PD-L1 status indeterminate, not evaluable, or missing: number analyzed (Participants) | 3 | 0 | 2
  Participants with baseline PD-L1 status indeterminate, not evaluable, or missing | 33.3 [0.8 to 90.6] |  | 0.0 [0.0 to 84.2]
  All randomized participants | 27.7 [22.9 to 32.9] | 47.4 [41.8 to 53.0] | 26.9 [22.1 to 32.0]

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose, up to 43 months
Groups:
- Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: Participants will receive treatment with nivolumab 3 mg/kg as a 30-minute infusion every 2 weeks and ipilimumab as a 30-minute infusion 1 mg/kg every 6 weeks.
- Nivolumab 240 mg + Chemotherapy: Participants will receive treatment with nivolumab 240 mg as a 30-minute infusion on Day 1 and Day 15, fluorouracil 800 mg/m²/day as an IV continuous infusion on Day 1 through Day 5 (for 5 days), and cisplatin 80 mg/m² as a 30- to 120-minute infusion on Day 1 of 4-week cycle.
- Chemotherapy: Participants will receive treatment with fluorouracil 800 mg/m²/day as an IV continuous infusion from Day 1 through Day 5 (for 5 days), and cisplatin 80 mg/m² as a 30- to 120-minute infusion on Day 1 of 4-week cycle.
Arm/Group | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Nivolumab 240 mg + Chemotherapy | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 215/322 | 200/310 | 224/304
Serious Adverse Events (participants affected / at risk) | 237/322 | 217/310 | 172/304
Other Adverse Events (participants affected / at risk) | 301/322 | 307/310 | 288/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=322) | Nivolumab 240 mg + Chemotherapy (N=310) | Chemotherapy (N=304)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 6 | 5
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 3
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 8 | 2 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 0
Hypophysitis (Endocrine disorders) | 6 | 0 | 0
Hypopituitarism (Endocrine disorders) | 6 | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 2 | 0 | 0
Thyroiditis (Endocrine disorders) | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1
Uveitis (Eye disorders) | 1 | 0 | 0
Vogt-Koyanagi-Harada disease (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Aorto-oesophageal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 4 | 5 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 12 | 20 | 16
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 1 | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 1 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 3
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Oesophageal mass (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 3 | 3 | 5
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 2 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 3 | 9 | 13
Oesophageal-pulmonary fistula (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagomediastinal fistula (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 5 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 2
Vomiting (Gastrointestinal disorders) | 4 | 4 | 12
Asthenia (General disorders) | 5 | 2 | 1
Catheter site discharge (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 2 | 0
Complication associated with device (General disorders) | 0 | 0 | 1
Death (General disorders) | 5 | 2 | 1
Disease progression (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 1
Feeling cold (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 2 | 1 | 1
Malaise (General disorders) | 2 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Nodule (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 1
Polyp (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 14 | 7 | 7
Sudden death (General disorders) | 1 | 2 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 9 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 2 | 3
Encephalitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 2 | 1
Large intestine infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Lung abscess (Infections and infestations) | 1 | 1 | 1
Lymph gland infection (Infections and infestations) | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Meningoencephalitis bacterial (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 31 | 33 | 20
Pneumonia bacterial (Infections and infestations) | 4 | 0 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 4 | 3 | 3
Septic shock (Infections and infestations) | 1 | 0 | 1
Stoma site cellulitis (Infections and infestations) | 1 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Atrio-oesophageal fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 5 | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stoma site extravasation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Adjusted calcium increased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 2 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Cortisol decreased (Investigations) | 1 | 0 | 0
Electrocardiogram Q wave abnormal (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 4 | 1
Platelet count decreased (Investigations) | 0 | 2 | 2
Transaminases increased (Investigations) | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 8 | 4 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 4 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4 | 4
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adult T-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 59 | 56 | 62
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0 | 0
Immune-mediated encephalopathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 1 | 0
Subdural hygroma (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1
Device leakage (Product Issues) | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Patient-device incompatibility (Product Issues) | 1 | 0 | 0
Assisted suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Pressure of speech (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 9 | 4
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Jejunostomy (Surgical and medical procedures) | 1 | 0 | 0
Oesophageal operation (Surgical and medical procedures) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Embolism (Vascular disorders) | 2 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 1
Internal haemorrhage (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Poor venous access (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 2
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=322) | Nivolumab 240 mg + Chemotherapy (N=310) | Chemotherapy (N=304)
Anaemia (Blood and lymphatic system disorders) | 82 | 151 | 107
Neutropenia (Blood and lymphatic system disorders) | 5 | 36 | 23
Hyperthyroidism (Endocrine disorders) | 20 | 7 | 1
Hypothyroidism (Endocrine disorders) | 44 | 21 | 1
Abdominal pain (Gastrointestinal disorders) | 22 | 22 | 18
Abdominal pain upper (Gastrointestinal disorders) | 16 | 20 | 13
Constipation (Gastrointestinal disorders) | 83 | 140 | 137
Diarrhoea (Gastrointestinal disorders) | 84 | 96 | 63
Dysphagia (Gastrointestinal disorders) | 35 | 39 | 30
Nausea (Gastrointestinal disorders) | 87 | 204 | 172
Stomatitis (Gastrointestinal disorders) | 33 | 99 | 75
Vomiting (Gastrointestinal disorders) | 52 | 74 | 60
Asthenia (General disorders) | 24 | 22 | 26
Fatigue (General disorders) | 53 | 82 | 63
Infusion site extravasation (General disorders) | 6 | 15 | 21
Malaise (General disorders) | 26 | 58 | 55
Mucosal inflammation (General disorders) | 5 | 36 | 30
Oedema peripheral (General disorders) | 31 | 45 | 25
Pyrexia (General disorders) | 76 | 62 | 48
Hepatic function abnormal (Hepatobiliary disorders) | 17 | 3 | 1
Pneumonia (Infections and infestations) | 35 | 31 | 29
Alanine aminotransferase increased (Investigations) | 45 | 26 | 13
Aspartate aminotransferase increased (Investigations) | 47 | 28 | 12
Blood alkaline phosphatase increased (Investigations) | 19 | 22 | 10
Blood creatinine increased (Investigations) | 12 | 42 | 39
Creatinine renal clearance decreased (Investigations) | 0 | 20 | 9
Lymphocyte count decreased (Investigations) | 8 | 16 | 9
Neutrophil count decreased (Investigations) | 10 | 75 | 61
Platelet count decreased (Investigations) | 12 | 46 | 36
Weight decreased (Investigations) | 41 | 40 | 35
Weight increased (Investigations) | 5 | 23 | 14
White blood cell count decreased (Investigations) | 12 | 58 | 41
Decreased appetite (Metabolism and nutrition disorders) | 69 | 160 | 155
Hypercalcaemia (Metabolism and nutrition disorders) | 12 | 20 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 20 | 22
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 | 25 | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 17 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 44 | 30
Hyponatraemia (Metabolism and nutrition disorders) | 31 | 54 | 36
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 17 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 18 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 10 | 16
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 14 | 19
Dizziness (Nervous system disorders) | 15 | 17 | 29
Dysgeusia (Nervous system disorders) | 10 | 23 | 19
Headache (Nervous system disorders) | 26 | 27 | 16
Neuropathy peripheral (Nervous system disorders) | 2 | 22 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 31 | 28
Insomnia (Psychiatric disorders) | 32 | 54 | 40
Renal impairment (Renal and urinary disorders) | 2 | 11 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 43 | 37
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 13 | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 12 | 53 | 63
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 | 19 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 42 | 42
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 13 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 59 | 37 | 19
Rash (Skin and subcutaneous tissue disorders) | 74 | 42 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 8 | 3
Hypertension (Vascular disorders) | 9 | 24 | 22
Hypotension (Vascular disorders) | 11 | 13 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT03143153/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT03143153/SAP_001.pdf